CLINICAL TRIAL: NCT03759717
Title: Molecular and Cellular Characterization of Skull Base Tumors
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Paul Gardner, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY19070185
Record Dates: First submitted 2018-10-31; First posted 2018-11-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Skull Base Neoplasm; Cellular Pathology
MeSH Terms: conditions — Skull Base Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Understanding the biology of skull base tumors will teach the investigators about the genesis and/or mechanisms of treatment resistance. The investigators hope to ultimately identify new targets which will add to the armamentarium by which to treat these tumors.

SUMMARY:
The purpose of the study is to analyze biological samples and genetic material for basic science research investigating the molecular and cellular characterization of skull base tumors.

DETAILED DESCRIPTION:
The overall goal of this proposal is to determine new molecular and cellular features that define tumor subtypes that are clinically actionable, may drive important changes in patient management, and/or elucidate novel chemotherapeutic options. Skull base tumors are currently diagnosed based on histopathologic criteria, on which post-operative management is based. However, the investigators hypothesize that each tumor type (eg. chordoma or chondrosarcoma) will have molecular and/or cellular subcategories that will redefine how to categorize and diagnose patients, predict clinical outcome, and optimally design a patient-specific management strategy. In addition, we aim to catalogue changes that occur after treatment after surgical resection, chemotherapy, and/or radiation by comparing primary and recurrent tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a skull base tumor

Exclusion Criteria:

* Insufficient tumor sample at time of resection

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a skull base tumor
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2028-10-03 (Estimated); Study Completion 2028-10-03 (Estimated)

PRIMARY OUTCOMES:
Patient overall survival will be measured and reported. | Through study completion, an average of 10 years
  There will be one outcome measure: overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gardner, MD, Principal Investigator — Associate Professor
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
If data is to be shared it will be de-identified with proper data use agreements in place.